CLINICAL TRIAL: NCT03115619
Title: A Multicenter, Post-Marketing, Non-Interventional, Observational Study to Evaluate Quality of Life in Patients in Greece With Idiopathic Pulmonary Fibrosis Under Treatment With Pirfenidone - The Pneumon Study
Brief Title: Quality of Life Study in Participants With IPF Under Pirfenidone Treatment
Acronym: PNEUMON
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39259
Record Dates: First submitted 2017-04-12; First posted 2017-04-14 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants With IPF: Observational data of participants with IPF under treatment with pirfenidone will be collected from the medical records as a part of their routine clinical visits at 12-week interval until study completion or early withdrawal (up to Week 52).
  Interventions: Drug: Pirfenidone

INTERVENTIONS:
Drug: Pirfenidone — Participants will receive pirfenidone therapy as per clinical practice or summary of product characteristics (SmPC).
  Other Names: Esbriet

SUMMARY:
This multicenter, post-marketing, observational study will evaluate quality of life in participants with Idiopathic Pulmonary Fibrosis (IPF) under treatment with pirfenidone (Esbriet).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants for whom pirfenidone has already been prescribed for IPF no more than 4 weeks prior to enrollment, according to their physicians' clinical decision and the terms in the SmPC

Exclusion Criteria:

* Participants who are participating in an interventional study or have received any investigational agent in the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in Greece with IPF under treatment with pirfenidone.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Quality of Life of Participants as Assessed by Saint George's Respiratory Questionnaire (SGQR) Score at the End of Treatment | Baseline, end of treatment (up to Week 52)

SECONDARY OUTCOMES:
Change From Baseline in Dyspnoea as Assessed by Medical Research Council (MRC) Breathlessness Scale Level at the End of Treatment | Baseline, end of treatment (up to Week 52)
Change From Baseline in Percent (%) Predicted Forced Vital Capacity (FVC) at the End of Treatment | Baseline, end of treatment (up to Week 52)
Change From Baseline in Annual FVC | From Baseline up to end of treatment (up to Week 52)
Change From Baseline in % Predicted Diffusing Lung Capacity for Carbon Monoxide (DLCO) at the End of Treatment | Baseline, end of treatment (up to Week 52)
Percentage of participants With Acute IPF Exacerbations, IPF-Related Death, Lung Transplant, or Respiratory-Related Hospitalization | from Baseline up to end of treatment (up to Week 52)
Percentage of Participants who are Compliant to Treatment | From Baseline up to end of treatment (up to Week 52)
  Treatment compliance will be assessed by the total number of dose reductions, dose interruptions, and the administered dosing intensity relative to the projected dose intensity during treatment.
Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interests | From Baseline up to end of treatment (up to Week 52)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Greece (7):
  - Sotiria Hospital for Diseases of the Chest, Academic Department of Pneumonology, Athens
  - University General Hospital of Athens "Attikon", B' University Pulmonary Clinic, Chaïdári
  - University General Hospital of Heraklio, Pulmonary Clinic, Heraklio
  - University General Hospital of Ioannina, Ioannina
  - General University Hospital of Larisa; Pneumonology Clinic, Larissa
  - General Hospital of Thessaloniki Papanikolaou; Uni Pneumonology Dept., Thessaloniki
  - Papanikolaou Hospital; Pneumonology Clinic, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided